CLINICAL TRIAL: NCT02122471
Title: A National, Randomized, 12-Week, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of Plecanatide (3.0 and 6.0 mg) in Patients With Chronic Idiopathic Constipation
Brief Title: 12-Week Study of Plecanatide for CIC (The National CIC3 Study)
Acronym: CIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP304203-03
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Chronic Idiopathic Constipation
Keywords: CIC; Constipation; Chronic Constipation; Synergy; Plecanatide
MeSH Terms: conditions — Constipation | interventions — plecanatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Plecanatide 3.0 mg (Experimental): Plecanatide tablets 3.0 mg QD for 12 weeks
  Interventions: Drug: Plecanatide
- Placebo (Placebo Comparator): Matching placebo tablets QD for 12 weeks
  Interventions: Drug: Placebo
- Plecanatide 6.0 mg (Experimental): Plecanatide tablets 6.0 mg QD for 12 weeks
  Interventions: Drug: Plecanatide

INTERVENTIONS:
Drug: Plecanatide
  Arms: Plecanatide 3.0 mg; Plecanatide 6.0 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to confirm that the investigational medication, plecanatide, is safe and effective in treating chronic idiopathic constipation.

DETAILED DESCRIPTION:
This is a national, randomized, 12-week, double-blind, placebo-controlled, study in approximately 1350 adult male and female patients with CIC comparing 2 doses of plecanatide to placebo. The study will be conducted at approximately 180 clinical study sites in the United States. The primary objective of the study is to evaluate the efficacy and safety of 3.0 and 6.0 mg of plecanatide administered once daily (QD) for 12 weeks in a population of patients with CIC. The study population will include only patients without other causes of constipation or other chronic conditions that could interfere with study assessments. Patients may not take laxatives (with the exception of the study-provided rescue medication, bisacodyl 5mg tablets), or a number of prohibited drugs that are known to cause constipation or diarrhea, during study participation.

There are 6 scheduled study visits, including the screening and follow-up visits. The planned duration of participation in this study will be 112 days and up to 155 days, with washout and all visit windows considered.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-80, inclusive
* Meets modified Rome III criteria for functional chronic idiopathic constipation for at least 3 months with symptom onset for at least 6 months
* Completed a colonoscopy in accordance with American Gastroenterological Association (AGA) colon cancer screening guidelines (5 years), with no clinically significant findings
* Willing to maintain a stable diet during the study

Exclusion Criteria:

* Loose stool (mushy) or watery (Bristol score 6 or 7) stool in the absence of any laxative or prohibited medicine for > 25% of Bowel Movements (BMs) during the 3 months prior to screening visit OR during the 14 day pre-treatment assessment
* Active peptic ulcer disease, diabetes or hypertension not adequately treated or not stable
* History of cathartic colon, laxative, enema abuse, or ischemic colitis
* Fecal impaction within 3 months of screening
* Patient has had /has any: diseases or conditions associated with constipation (GI or CNS), structural abnormality of the GI tract or gastric bypass surgery, pelvic floor dysfunction, pseudo-obstruction, active infectious gastritis, diverticulitis, anal fissures or any disease or condition that can affect GI motility or defecation or can be associated with abdominal pain
* Unexplained and clinically significant "alarm symptoms" including lower GI bleeding, iron-deficiency anemia, weight loss or systemic signs of infection or colitis
* Major surgery, stroke or myocardial infarction (MI) within 60 days of screening
* Participated in a previous plecanatide clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1410 (Actual)
Dates: Start 2014-04; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Layton, Study Director — Synergy Pharmaceuticals Inc.
Locations (122):
- United States (122):
  - Synergy Research Site, Anniston, Alabama
  - Synergy Research Site, Huntsville, Alabama
  - Synergy Research Site, Chandler, Arizona
  - Synergy Research Site, Goodyear, Arizona
  - Synergy Research Site, Tucson, Arizona
  - Synergy Research Site, Anaheim, California
  - Synergy Research Site, Artesia, California
  - Synergy Research Site, Carmichael, California
  - Synergy Research Site, Corona, California
  - Synergy Research Site, Encino, California
  - Synergy Research Site, Garden Grove, California
  - Synergy Research Site, Glendale, California
  - Synergy Research Site, La Mirada, California
  - Synergy Research Site, Laguna Hills, California
  - Synergy Research Site, Los Angeles, California
  - Synergy Research Site, Newport Beach, California
  - Synergy Research Site, Oceanside, California
  - Synergy Research Site, Orange, California
  - Synergy Research Site, Sacramento, California
  - Synergy Research Site, San Bernardino, California
  - Synergy Research Site, San Diego, California
  - Synergy Research Site, Upland, California
  - Synergy Research Site, Ventura, California
  - Synergy Research Site, Denver, Colorado
  - Synergy Research Site, Littleton, Colorado
  - Synergy Research Site, Stamford, Connecticut
  - Synergy Research Site, Aventura, Florida
  - Synergy Research Site, Boynton Beach, Florida
  - Synergy Research Site, Bradenton, Florida
  - Synergy Research Site, Brandon, Florida
  - Synergy Research Site, Brooksville, Florida
  - Synergy Research Site, Clearwater, Florida
  - Synergy Research Site, DeLand, Florida
  - Synergy Research Site, Fort Lauderdale, Florida
  - Synergy Research Site, Gainesville, Florida
  - Synergy Research Site, Hialeah, Florida
  - Synergy Research Site, Hollywood, Florida
  - Synergy Research Site, Homestead, Florida
  - Synergy Research Site, Jacksonville, Florida
  - Synergy Research Site, Miami, Florida
  - Synergy Research Site, Miami Lakes, Florida
  - Synergy Research Site, Miami Springs, Florida
  - Synergy Research Site, New Port Richey, Florida
  - Synergy Research Site, North Miami Beach, Florida
  - Synergy Research Site, Orlando, Florida
  - Synergy Research Site, Ormond Beach, Florida
  - Synergy Research Site, Pembroke Pines, Florida
  - Synergy Research Site, Plant City, Florida
  - Synergy Research Site, Plantation, Florida
  - Synergy Research Site, Saint Cloud, Florida
  - Synergy Research Site, Sarasota, Florida
  - Synergy Research Site, Seminole, Florida
  - Synergy Research Site, St. Petersburg, Florida
  - Synergy Research Site, Tamarac, Florida
  - Synergy Research Site, Tampa, Florida
  - Synergy Research Site, West Palm Beach, Florida
  - Synergy Research Site, Atlanta, Georgia
  - Synergy Research Site, Savannah, Georgia
  - Synergy Research Site, Snellville, Georgia
  - Synergy Research Site, Blackfoot, Idaho
  - Synergy Research Site, Boise, Idaho
  - Synergy Research Site, Chicago, Illinois
  - Synergy Research Site, Oak Lawn, Illinois
  - Synergy Research Site, Schaumburg, Illinois
  - Synergy Research Site, Evansville, Indiana
  - Synergy Research Site, Madisonville, Kentucky
  - Synergy Research Site, Owensboro, Kentucky
  - Synergy Research Site, Monroe, Louisiana
  - Synergy Research Site, Shreveport, Louisiana
  - Synergy Research Site, Columbia, Maryland
  - Synergy Research Site, Watertown, Massachusetts
  - Synergy Research Site, Buckley, Michigan
  - Synergy Research Site, St Louis, Missouri
  - Synergy Research Site, Omaha, Nebraska
  - Synergy Research Site, Las Vegas, Nevada
  - Synergy Research Site, Stateline, Nevada
  - Synergy Research Site, Newington, New Hampshire
  - Synergy Research Site, Blackwood, New Jersey
  - Synergy Research Site, Albuquerque, New Mexico
  - Synergy Research Site, Elmsford, New York
  - Synergy Research Site, New Hyde Park, New York
  - Synergy Research Site, New York, New York
  - Synergy Research Site, Cary, North Carolina
  - Synergy Research Site, Concord, North Carolina
  - Synergy Research Site, Hickory, North Carolina
  - Synergy Research Site, High Point, North Carolina
  - Synergy Research Site, Raleigh, North Carolina
  - Synergy Research Site, Cincinnati, Ohio
  - Synergy Research Site, Cleveland, Ohio
  - Synergy Research Site, Columbus, Ohio
  - Synergy Research Site, Kettering, Ohio
  - Synergy Research Site, Middleburg Heights, Ohio
  - Synergy Research Site, Sylvania, Ohio
  - Synergy Research Site, Wadsworth, Ohio
  - Synergy Research Site, Oklahoma City, Oklahoma
  - Synergy Research Site, Jenkintown, Pennsylvania
  - Synergy Research Site, Levittown, Pennsylvania
  - Synergy Research Site, Pittsburgh, Pennsylvania
  - Synergy Research Site, Upper Saint Clair, Pennsylvania
  - Synergy Research Site, Greer, South Carolina
  - Synergy Research Site, Moncks Corner, South Carolina
  - Synergy Research Site, Bristol, Tennessee
  - Synergy Research Site, Franklin, Tennessee
  - Synergy Research Site, Jefferson City, Tennessee
  - Synergy Research Site, Kingsport, Tennessee
  - Synergy Research Site, Knoxville, Tennessee
  - Synergy Research Site, Memphis, Tennessee
  - Synergy Research Site, Nashville, Tennessee
  - Synergy Research Site, Arlington, Texas
  - Synergy Research Site, Austin, Texas
  - Synergy Research Site, Carrollton, Texas
  - Synergy Research Site, Channelview, Texas
  - Synergy Research Site, Dallas, Texas
  - Synergy Research Site, Gonzales, Texas
  - Synergy Research Site, Houston, Texas
  - Synergy Research Site, Pharr, Texas
  - Synergy Research Site, Plano, Texas
  - Synergy Research Site, San Antonio, Texas
  - Synergy Research Site, Draper, Utah
  - Synergy Research Site, Newport News, Virginia
  - Synergy Research Site, Sterling, Virginia
  - Synergy Research Site, Richland, Washington

REFERENCES:
- [Derived] Cash BD, Sharma A, Walker A, Laitman AP, Chang L. Plecanatide for the treatment of chronic idiopathic constipation and irritable bowel syndrome with constipation: Post hoc analyses of placebo-controlled trials in adults with severe constipation. Neurogastroenterol Motil. 2023 Sep;35(9):e14632. doi: 10.1111/nmo.14632. Epub 2023 Jun 18. PMID 37332239
- [Derived] Moshiree B, Schoenfeld P, Franklin H, Rezaie A. The Effect of Acid Suppression Therapy on the Safety and Efficacy of Plecanatide: Analysis of Randomized Phase III Trials. Clin Ther. 2022 Jan;44(1):98-110.e1. doi: 10.1016/j.clinthera.2021.11.009. Epub 2022 Jan 25. PMID 35086735
- [Derived] Menees SB, Franklin H, Chey WD. Evaluation of Plecanatide for the Treatment of Chronic Idiopathic Constipation and Irritable Bowel Syndrome With Constipation in Patients 65 Years or Older. Clin Ther. 2020 Jul;42(7):1406-1414.e4. doi: 10.1016/j.clinthera.2020.05.012. Epub 2020 Jul 10. PMID 32660770
- [Derived] DeMicco M, Barrow L, Hickey B, Shailubhai K, Griffin P. Randomized clinical trial: efficacy and safety of plecanatide in the treatment of chronic idiopathic constipation. Therap Adv Gastroenterol. 2017 Nov;10(11):837-851. doi: 10.1177/1756283X17734697. Epub 2017 Oct 25. PMID 29147135

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The data are correct and approved in the NDA. 1410 randomized subj.including 95 (index and non-index) duplicate subj. The index subj (22) were duplicate appeared the first time in the study and the same subject appeared in other studies or sites were non-index duplicate (73) who were excluded in the ITT population (1337).
Groups:
- Plecanatide 3 mg: Plecanatide tablets 3 mg QD for 12 weeks
- Plecanatide 6 mg: Plecanatide tablets 6 mg QD for 12 weeks
Period: Overall Study
Arm/Group | Placebo | Plecanatide 3 mg | Plecanatide 6 mg
Started | 445 | 443 | 449
Completed | 406 | 392 | 405
Not Completed | 39 | 51 | 44

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Plecanatide 3 mg | Plecanatide 6 mg | Total
Number analyzed (Participants) | 445 | 443 | 449 | 1337
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (14.59) | 45.5 (14.38) | 45.3 (14.47) | 45.1 (14.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 350 | 345 | 353 | 1048
  Male | 95 | 98 | 96 | 289

OUTCOME MEASURES:

1. Primary Outcome: Number of Durable Overall CSBM Responders, Mean Replacement Approach
Description: The primary efficacy endpoint was measured by the number of durable overall CSBM responders over the 12-week Treatment Period. A durable overall CSBM responder was defined as a weekly CSBM responder for at least 9 of the 12 treatment weeks, including at least 3 of the last 4 weeks. A CSBM weekly responder was defined as a patient who has ≥ 3 Complete Spontaneous Bowel Movements (CSBMs) per week and an increase from baseline of ≥1 CSBM for that week. A CSBM was a bowel movement that occurred in the absence of laxative use within 24 hours and was associated with the feeling of complete evacuation.
Time Frame: 12-Week Treatment Period
Population: The modified ITT population (1310 subjects) for primary outcome was ITT population minus 27 subjects eliminated from two OAI sites. The ITT population (1337) as described in the Participate Flow consisted of the randomized subjects (1410) excluding 73 non-index subjects. "Index" subjects were duplicate subjects appeared once in the ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Plecanatide 3 mg | Plecanatide 6 mg
Number analyzed (Participants) | 440 | 430 | 440
Participants | 57 | 88 | 88

2. Secondary Outcome: Change From Baseline in CSBMs (CSBMs/Week) Over the 12-week Treatment Period , Mean Replacement Approach
Description: The change from baseline in the number of Complete Spontaneous Bowel Movements (CSBMs) over the 12-week Treatment Period was analyzed. Baseline was the mean number of CSBMs recorded during the 2-week baseline diary assessment period prior to the first dose of study drug. A CSBM was a bowel movement that occurred in the absence of laxative use within 24 hours and was associated with the feeling of complete evacuation.
Time Frame: Baseline and 12 weeks
Population: A total of 1288 patients included in ITT-E population for secondary outcome which consisted of the randomized subjects (1410) excluding 95 duplicate subjects as described in the Participate Flow and 27 subjects eliminated from two OAI sites.
Measure: Least Squares Mean (Standard Error); unit: CSBMs per week
Groups:
- Plecanatide 6 mg: Plecanatide tablets 6 mg QD for 12 week
Arm/Group | Placebo | Plecanatide 3 mg | Plecanatide 6 mg
Number analyzed (Participants) | 432 | 422 | 434
CSBMs per week
  Baseline | 1.41 (0.138) | 2.34 (0.139) | 2.19 (0.138)
  12 weeks | 1.69 (0.159) | 2.66 (0.162) | 2.50 (0.159)

3. Secondary Outcome: Change From Baseline in SBMs (SBMs/Week) Over the 12-week Treatment Period, Mean Replacement Approach
Description: The change from baseline in the number of Spontaneous Bowel Movement (SBM) over the 12-week Treatment Period was analyzed. Baseline was the mean number of SBMs recorded during the 2-week baseline diary assessment period prior to the first dose of study drug. The weekly SBM totals were derived from the daily diary entries reported during the Treatment Period.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SBMs per week
Arm/Group | Placebo | Plecanatide 3 mg | Plecanatide 6 mg
Number analyzed (Participants) | 432 | 422 | 434
SBMs per week
  Baseline | 1.55 (1.591) | 1.79 (2.084) | 1.63 (1.673)
  12 weeks | 1.81 (2.879) | 3.25 (3.938) | 3.10 (4.164)

4. Secondary Outcome: Change From Baseline in Average Weekly SBM Stool Consistency Over the 12-week Treatment Period, Mean Replacement Approach
Description: The change from baseline in the stool consistency score (i.e. BSFS) over the 12-week Treatment Period was analyzed. Baseline was the mean BSFS score recorded during the 2-week baseline diary assessment period prior to the first dose of study drug. The weekly mean BSFS score per patient was derived from the BSFS entries reported during the Treatment Period in the Daily Symptom Diary.
  The stool consistency of each bowel movement (BM) was assessed by patients using the 7-point Bristol Stool Form Scale [BSFS] from 1 to 7.
  1. = separate hard lumps like nuts (difficult to pass)
  2. = sausage shaped but lumpy
  3. = like a sausage but with cracks on its surface
  4. = like a sausage or snake, smooth and soft
  5. = soft blobs with clear-cut edges (passed easily)
  6. = fluffy pieces with ragged edges, a mushy stool
  7. = watery, no solid pieces (entirely liquid)
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Plecanatide 3 mg | Plecanatide 6 mg
Number analyzed (Participants) | 432 | 422 | 434
score on a scale
  Baseline | 2.35 (1.090) | 2.16 (1.036) | 2.27 (1.113)
  12 weeks | 1.02 (1.346) | 1.71 (1.475) | 1.59 (1.497)

5. Secondary Outcome: Change From Baseline in Average Weekly Straining Score Over the 12-week Treatment Period, Mean Replacement Approach
Description: The change from baseline in the straining score over the 12-week Treatment Period was analyzed. Baseline was the mean of non-missing straining scores recorded during the 2-week baseline diary assessment period prior to the first dose of study drug. The weekly average straining score was derived from the straining scores reported during the Treatment Period in the Daily Symptom Diary. The severity of straining during bowel movements was assessed on a 5-point Likert scale where 0 = none, 1 = mild, 2 = moderate, 3 = severe, and 4 = very severe.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Plecanatide 3 mg | Plecanatide 6 mg
Number analyzed (Participants) | 432 | 422 | 434
score on a scale
  Baseline | 2.42 (0.855) | 2.46 (0.859) | 2.47 (0.888)
  12 weeks | -0.79 (1.132) | -1.09 (1.092) | -1.04 (1.084)

ADVERSE EVENTS:
Description: The data are correct and approved in the NDA. The ITT-S population (1402) was more than the ITT population (1337) in the Participant Flow because all duplicate subjects (index and non-index) who received at lease one dose of study drug were included in the ITT-S population. A total of 1410 randomized subjects, of which eight subjects were not treated with the study drug after being enrolled and resulted in 1402 subjects.
Arm/Group | Placebo | Plecanatide 3 mg | Plecanatide 6 mg
Serious Adverse Events (participants affected / at risk) | 8/466 | 8/467 | 4/469
Other Adverse Events (participants affected / at risk) | 15/466 | 25/467 | 31/469
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=466) | Plecanatide 3 mg (N=467) | Plecanatide 6 mg (N=469)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (2) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=466) | Plecanatide 3 mg (N=467) | Plecanatide 6 mg (N=469)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 15 (15) | 21 (25)
Headache (Nervous system disorders) | 9 (10) | 10 (10) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes